CLINICAL TRIAL: NCT03693443
Title: Oral Health Beliefs, Knowledge, and Behavioral Attitudes of Egyptian Mothers Towards Early Childhood Caries
Brief Title: Knowledge and Behavior Toward Early Childhood Caries
Status: Completed | Type: Observational
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Naglaa Ibrahim Ezz, Lecturer, October University for Modern Sciences and Arts
Other Study IDs: ETH6
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-12

CONDITIONS: Early Childhood Caries
Keywords: knowledge; behaviors; Early childhood caries
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: early childhood caries — a questionnaire evaluates the oral health beliefs, knowledge, and behaviors of a sample representing Egyptian mothers toward early childhood caries

SUMMARY:
400 mothers are at least 18 years of age who have at least a child with minimum age of 6 years or even younger will be selected from the outpatient clinics of October University for Modern Sciences and arts (MSA). The questionnaire will be administrated to obtain socio demographic information and to assess their oral health beliefs, knowledge, behaviors and the possible barriers for their accessing oral health care.

ELIGIBILITY:
Inclusion Criteria:

* mothers are at least 18 years of age who have at least a child with minimum age of 6 years or even younger

Exclusion Criteria:

* mothers are refuse to participate in the study or sign the consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Mothers are at least 18 years of age who have at least a child with minimum age of 6 years or even younger will be selected from the outpatient clinics of October University for Modern Sciences and arts, Cairo city, the capital of Egypt.
Sampling Method: Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
evaluation of the oral health beliefs, knowledge, and behavioral attitudes towards early childhood caries | 3 months
  data collected from the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa I Ezz El Din, lecturer, Principal Investigator — October University for Modern Sciences and Arts
Locations (1):
- October University of Modern Sciences and Arts, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No